CLINICAL TRIAL: NCT04395963
Title: Leader's Eye Tracking Patterns Changes During High Fidelity Simulation Scenarios of Postpartum Hemorrhage
Brief Title: Eye Tracking and Simulated Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Other Study IDs: EESOA7
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Simulation of Physical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tobii Pro Glasses 50 Hz wearable wireless eye tracker — This system can measure eye movements using cameras integrated into the eyeglasses which record the corneal reflection of infrared lighting to track pupil position, mapping the subject's focus of attention on video recordings of the subject's field of vision (gaze).

SUMMARY:
Eye tracking is the process of measuring an individual's eye movements in order to reflect their attentional behavior by using a device called an eye- tracker.

This study uses eye-tracking methodology to observe the gaze patterns of participants to a high fidelity simulation scenario of postpartum hemorrhage acting in the role of leader to evaluate the relationship between eye-tracking patterns and leadership and team behavioral and technical skills.

DETAILED DESCRIPTION:
This study will include 5 groups of anesthesia trainees consisting of 5 participants each. Each group will practice a standardized high-fidelity scenario on postpartum hemorrhage (PPH) which will be repeated for four times. All the scenarios will be video recorded.

All groups will receive a technical briefing on the PPH guidelines before the scenario, and after having assigned to each participant a role (leader anesthesiologist, junior anesthesiologist, obstetrician, and midwife) they will practice a standardized 15 minutes scenario with a high fidelity manikin. A debriefing with an expert debriefer will be performed after each scenario.

The participant acting as the leader will practice the scenario while wearing a pair of eye-tracking glasses (Tobii Pro Glasses 50 Hz wearable wireless eye-tracker). All the eye-tracking video-recordings will be stored and analyzed by using a Tobii Pro Lab Software. Specific areas of interest (AOI), to define regions of a displayed stimulus, and to extract metrics specifically for those regions will be selected. Number and duration of fixations, visit counts and their duration for each area of interest and for each scenario will be examined. Eye-tracking metrics will be mapped as gaze plots and heat maps. Two independent observers will review the scenario video recordings and will assing a score to the leader and team behavioral and technical skills. These scores will be correlated to eye tracking metrics.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia trainee

Exclusion Criteria:

* severe vision defects

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: anesthesia trainee
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Eye-tracking and behavioral scores | 15 minutes
  Correlation between eye-traking metrics, leader's behavior and team efficacy during the scenario

SECONDARY OUTCOMES:
Eye-tracking and behavioral scores during the learning process | 15 minutes
  Correlation between eye-traking metrics, leader's behavior and team efficacy during the scenario and differences between the different scenarios played over the time

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Eesoa Simulation Center, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tien T, Pucher PH, Sodergren MH, Sriskandarajah K, Yang GZ, Darzi A. Eye tracking for skills assessment and training: a systematic review. J Surg Res. 2014 Sep;191(1):169-78. doi: 10.1016/j.jss.2014.04.032. Epub 2014 Apr 24. PMID 24881471
- [Derived] Capogna E, Capogna G, Raccis D, Salvi F, Velardo M, Del Vecchio A. Eye tracking metrics and leader's behavioral performance during a post-partum hemorrhage high-fidelity simulated scenario. Adv Simul (Lond). 2021 Feb 4;6(1):4. doi: 10.1186/s41077-021-00156-2. PMID 33541439